CLINICAL TRIAL: NCT03849586
Title: Prospective Registry for Patients Undergoing Penile Prosthesis Implantation for Male Erectile Dysfunction
Brief Title: Registry for Patients Undergoing Penile Prosthesis Implantation for Male Erectile Dysfunction
Acronym: PHOENIX
Status: Active, not recruiting | Type: Observational
Sponsor: European Association of Urology Research Foundation (Other)
Collaborators: Boston Scientific Corporation (Industry); Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: EAU-RF 2018-01
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Erectile Dysfunction
Keywords: penile prosthesis implant
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective collection of pre-defined parameters on the surgical treatment of male erectile dysfunction using Penile Prosthesis Implants (PPIs).

DETAILED DESCRIPTION:
This will be a prospective collection of pre-defined parameters on the surgical treatment of male erectile dysfunction using Penile Prosthesis Implants (PPIs). The data collection will be undertaken from multiple centres in Europe. The participation will be by open invitation from the European Association of Urology (EAU) Section of Genitourinary Reconstructive Surgeons (ESGURS) to all its members, along with other urologists undertaking these procedures.

There will be no restriction on the number of patients enrolled per centre as long as they are consecutive. The aim is to have a long term collection of the dataset from as many centres as possible. An initial assessment for the robustness of the data collection and first clinical evaluation of the data collected will be performed 1 and 2 years after recruitment of the first patient by a nominated steering committee. Thereafter, the evaluations will be performed every 2 years until the end of Registry (10 years after the first patient was enrolled).

ELIGIBILITY:
Inclusion Criteria:

* Male patient undergoing a surgical penile prosthesis implant for treatment of erectile dysfunction.
* Participant is willing and able to give informed consent for participation in the Registry and is able to complete the questionnaires.

Exclusion Criteria:

* Participating center is unable to contribute consecutive patients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients undergoing a surgical Penile Prosthesis Implant for treatment of erectile dysfunction.
Sampling Method: Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2032-02 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction score | at week 12, year 1, 2, 4, 6, 8 and 10 after surgery
  Patient Satisfaction score is defined as the mean patient satisfaction score as indicated by the Modified Patient EDITS Questionnaire. All items on the Patient EDITS will be scored from zero (no satisfaction or dissatisfaction) to four (high satisfaction). The mean satisfaction score for each patient will be calculated. To place scores in an easily interpretable metric, each mean score will be multiplied by 25 so that EDITS scores could range from a low of 0 (extremely low treatment satisfaction) to a high of 100 extremely high treatment satisfaction).

SECONDARY OUTCOMES:
Partner Satisfaction score | at week 12, year 1, 2, 4, 6, 8 and 10 after surgery
  Partner Satisfaction score is defined as the mean partner satisfaction score as indicated by the Modified Partner EDITS Questionnaire. All items on the Partner EDITS will be scored from zero (no satisfaction or dissatisfaction) to four (high satisfaction). The mean satisfaction score for the partner will be calculated. To place scores in an easily interpretable metric, each mean score will be multiplied by 25 so that EDITS scores could range from a low of 0 (extremely low treatment satisfaction) to a high of 100 extremely high treatment satisfaction).
Patient satisfaction rate | at week 12, year 1, 2, 4, 6, 8 and 10 after surgery
  The number of patients with an EDITS score ≥ 50 compared to the total number of patients
Partner satisfaction rate | at week 12, year 1, 2, 4, 6, 8 and 10 after surgery
  The number of partners with an EDITS score ≥ 50 compared to the total number of partners
Overall time being satisfied with treatment since implantation | up to 10 years post surgery
  The interval from the date of regaining a patient EDITS score of 50 or more until the time of EDITS score of less than 50
International Index of Erectile Function - 5 (IIEF short form/SHIM) questionnaire | at baseline, week 12, year 1, 2, 4, 6, 8 and 10 after surgery
  The IIEF-5 score is the sum of the ordinal responses to five items; thus, the score can range from 0 to 25. Erectile Dysfunction (ED) severity can be classified into the following five categories based on IIEF-5 scores; severe (0-7), moderate (8-11), mild to moderate (12-16), mild (17-21), and no ED (22- 25). Mean IIEF-5 scores will be calculated at the indicated time points and numbers / percentages of patients in the different ED severity categories. Also change in IIEF-5 score compared to baseline will be calculated.
Sexual Encounter Profile (SEP) questions 2 and 3 | at baseline, week 12, year 1, 2, 4, 6, 8 and 10 after surgery
  For SEP question 2 and 3, scores are percentage of yes responses relative to number of sexual attempts/encounters. Proportions of yes responses will be treated as continuous variables. Post-operative results will also be compared to baseline.
EQ-5D-5L quality of life questionnaire | at baseline, week 12, year 1, 2, 4, 6, 8 and 10 after surgery
  Results of the EQ-5D-5L quality of life questionnaire will be analyzed as described in the EuroQol EQ-5D-5L user guide. Post-operative results will also be compared to baseline.
Quality of Life and Sexuality with Penile Prosthesis (QoLSPP) questionnaire | at week 12, year 1, 2, 4, 6, 8 and 10 after surgery
  QoLSPP is a 16-item questionnaire, with 4 domains: the functional, relational, social and personal domain. Responses are structured according to a six-point Likert scale, in most cases ranging from "never" (0) to "always" (5), where higher values represent more positive responses. Individual item scores will be analyzed as well as domain scores.
Complications | during surgery and up to 10 years after surgery
  Type of complications, associated symptoms and whether or not a revision was needed will be recorded.
Immediate Postoperative complications | until 2 weeks after surgery
  Type of complications, associated symptoms and whether or not a revision was needed will be recorded and classified according to the Clavien Dindo grading system.
Time of first activation, first cycling, first use, first intercourse, first orgasm, if applicable | up to 10 years post surgery
  The date of first cycling (inflating and deflating the prosthesis several times), the date of first activation and first use for sexual activity, the date of first sexual intercourse and the date of first orgasm, if applicable, will be reported.
Time being revision-free | up to 10 years post surgery
  The interval from the date of surgery to the date of revision whereby revision is defined as any urogenital surgical intervention that is related to the function, placement, or site reaction to the implanted device
Revision-free rate | at 1, 2, 4, 6, 8 and 10 years of Registry follow-up
  The number of patients who are revision-free compared to the total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Koen van Renterghem, MD, PhD, Principal Investigator — Jessa Hospital, Hasselt, Belgium
Locations (30):
- Belgium (5):
  - University Hospital Antwerp, Antwerp
  - AZ Sint-Jan, Bruges
  - AZ Maria Middelares, Ghent
  - Jessa Hospital, Hasselt
  - UZ Leuven, Leuven
- CHU Lyon Sud, Lyon, France
- Germany (2):
  - University Hospital Essen (AöR), Essen
  - University Hospital Schleswig Holstein, Lübeck
- Italy (3):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - Azienda Ospedaliero-Universitaria "Ospedali Riuniti" di Foggia, Foggia
  - Casa di Cura Città di Parma, Parma
- Centro Hospitalar Universitario Lisboa Norte, Lisbon, Portugal
- Spain (14):
  - Fundació Puigvert, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario HM Montepríncipe, Boadilla del Monte
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Zarzuela, Madrid
  - Lyx Institute of Urology, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Rey Juan Carlos, Móstoles
  - Instituto Médico Rosselló, Palma de Mallorca
  - Marques de Valdecilla University Hospital, Santander
- Sweden (2):
  - Lund University, Skane Hospital,, Malmo
  - Karolinska University Hospital, Stockholm
- United Kingdom (2):
  - St.George's University Hospital, London
  - UCLH, London

IPD SHARING:
Plan to Share IPD: Undecided
Investigators may share anonymized individual data with residents/urologist interested to analyze and publish the results of the registry

REFERENCES:
- [Background] van Renterghem K, Deho F. Perspective on the PHOENIX trial: prospective registry for patients undergoing penile prosthesis implantation for male erectile dysfunction in multiple European centers. Int J Impot Res. 2023 Jun;35(4):329-331. doi: 10.1038/s41443-022-00547-7. Epub 2022 Feb 26. No abstract available. PMID 35220417
- [Result] van Renterghem K, Jorissen C, Van Huele A. Penile length changes after penile implant surgery. J Sex Med. 2023 Nov 30;20(12):1364-1366. doi: 10.1093/jsxmed/qdad125. No abstract available. PMID 38037429
- [Result] Van Renterghem K, De Bruyn H, Yebes A, Calopedos R, Deho F, Torremade J, D'Anna M, Bettocchi C, Gomez BG, Caris C, Witjes W, Moncada I, Ralph D; EAU Research Foundation PHOENIX Study Group. Early complications after penile prosthesis surgery: findings from the PHOENIX multicenter registry. Int J Impot Res. 2025 May 7. doi: 10.1038/s41443-025-01080-z. Online ahead of print. PMID 40335744
- See also: EAU Research Foundation website — https://uroweb.org/research/projects/